CLINICAL TRIAL: NCT00248781
Title: Home-based Exercise Via a Telecommunications System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: E2777-R
Record Dates: First submitted 2005-11-02; First posted 2005-11-04 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2013-12

CONDITIONS: Functional Limitation
Keywords: Activities of daily living; Aging; Exercise; Weight lifting
MeSH Terms: conditions — Motor Activity

ARMS (2):
- Arm 1 (Experimental): exercise
  Interventions: Device: Telecommunications system
- Arm 2 (Other): health education
  Interventions: Device: attention control

INTERVENTIONS:
Device: Telecommunications system
  Arms: Arm 1
Device: attention control — health education
  Arms: Arm 2

SUMMARY:
This study is investigating the effects of a home-based resistance exercise program, administered via an interactive telecommunications system, in functionally limited older veterans.

DETAILED DESCRIPTION:
Inactivity and a sedentary lifestyle have been shown to accelerate and exaggerate the age-related decline in muscle strength. In this context, a rapid decline in strength among older adults has been linked to physical frailty, falls, functional decline, impaired mobility, and nursing home placement. Substantial evidence now suggests that habitual physical activity is associated with the maintenance of muscle strength and physical function well into the 8th and 9th decades of life. We propose to investigate the effects of a home-based resistance exercise program, administered via an interactive telecommunications system without the participation of health professionals, in functionally limited older veterans. Subjects will be randomized to either the automated exercise group or an attention placebo control group. The exercise group will undergo resistance training at home three times a week for 6 months, guided by the telecommunications system, followed by a 6-month maintenance phase of less frequent interaction with the system. Outcome measurements will include muscle strength and physical performance related to daily activities at 3, 6, and 12 months to determine the efficacy of the intervention and the time course and durability of the effect. The control group will also interact with the telecommunications system once a week for the whole year, but no exercise will be prescribed. If this home-based, automated, interactive exercise program is effective, it will provide a low-cost easily disseminated approach to improving the strength and functional status of older veterans

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years
* Ability to use a telephone without assistance

Exclusion Criteria:

* Angina pectoris
* Myocardial infarction
* Ventricular dysrhythmia currently receiving therapy
* Systolic blood pressure 165 mm Hg or diastolic blood pressure 100 mm Hg

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 103 (Actual)
Dates: Start 2003-09; Primary Completion 2009-04 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David William Sparrow, DSc, Principal Investigator — VA Boston Health Care System
Locations (1):
- VA Boston Health Care System, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Automated Exercise Group: Telecommunications system for exercise
- Attention Control Group: attention control (health education)
Period: Overall Study
Arm/Group | Automated Exercise Group | Attention Control Group
Started | 52 | 51
Completed | 42 | 47
Not Completed | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Telecommunications system for exercise
- Arm 2: attention control (health education)
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (7.5) | 71.7 (7.2) | 71 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 35 | 36 | 71
Region of Enrollment [Number; unit: participants]
  United States | 52 | 51 | 103

OUTCOME MEASURES:

1. Primary Outcome: Knee Extension Strength
Description: The peak force measured during the bilateral knee extension exercise against the highest level of a hydraulic resistance system
Time Frame: 6 months
Population: number of subjects completing 6 month evaluations
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Automated Exercise Group | Attention Control Group
Number analyzed (Participants) | 45 | 48
kg | 20.4 (0.59) | 19.5 (0.65)

2. Secondary Outcome: Knee Extension Strength (Durability)
Description: as for outcome 1
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Automated Exercise Group | Attention Control Group
Number analyzed (Participants) | 42 | 47
kg | 20.3 (0.71) | 19.4 (0.66)

3. Primary Outcome: Knee Flexion Strength
Description: The peak force measured during the bilateral knee flexion exercise against the highest level of a hydraulic resistance system
Time Frame: 6 months
Population: Number of subjects completing 6 month evaluations
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Automated Exercise Group | Attention Control Group
Number analyzed (Participants) | 45 | 48
kg | 34.3 (0.76) | 32.2 (0.77)

4. Primary Outcome: Single Leg Stance With Eyes Open
Description: Length of time standing on one leg without moving the support foot, touching the floor or support leg with suspended foot, or requiring assistance.
Time Frame: 6 months
Population: The number of subjects completing 6 month evaluations
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Automated Exercise Group | Attention Control Group
Number analyzed (Participants) | 45 | 48
s | 20.9 (1.30) | 17.4 (1.30)

5. Primary Outcome: Tandem Stance
Description: Length of time standing with the heel of one foot touching the toe of the other foot keeping the feet in a straight line.
Time Frame: 6 months
Population: The number of subjects completing 6 month evaluations
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Automated Exercise Group | Attention Control Group
Number analyzed (Participants) | 45 | 48
s | 54.8 (1.9) | 50.5 (2.35)

6. Primary Outcome: Six-minute Walk
Description: Total distance walked during 6 minutes. Subjects were instructed to walk up and down a 100-foot level hallway as far as they could in 6 minutes.
Time Frame: 6 months
Population: The number of subjects completing 6 month evaluations
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Automated Exercise Group | Attention Control Group
Number analyzed (Participants) | 45 | 48
m | 450.6 (5.09) | 449.8 (5.22)

7. Secondary Outcome: Knee Flexion Strength (Durability)
Description: as for outcome 3
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Automated Exercise Group | Attention Control Group
Number analyzed (Participants) | 42 | 47
kg | 34.5 (0.81) | 32.5 (0.82)

8. Secondary Outcome: Single Leg Stance With Eyes Open (Durability)
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Automated Exercise Group | Attention Control Group
Number analyzed (Participants) | 42 | 47
s | 20.1 (1.35) | 16.6 (1.39)

9. Secondary Outcome: Tandem Stance (Durability)
Description: as for outcome 5
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Automated Exercise Group | Attention Control Group
Number analyzed (Participants) | 42 | 47
s | 55.8 (2.18) | 51.6 (2.38)

10. Secondary Outcome: Six-minute Walk (Durability)
Description: as for outcome 6
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Automated Exercise Group | Attention Control Group
Number analyzed (Participants) | 42 | 47
m | 446.8 (4.77) | 446.1 (4.91)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Automated Exercise Group | Attention Control Group
Serious Adverse Events (participants affected / at risk) | 6/52 | 7/51
Other Adverse Events (participants affected / at risk) | 8/52 | 7/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Automated Exercise Group (N=52) | Attention Control Group (N=51)
stroke (Cardiac disorders) | 1 (1) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
bypass surgery (Cardiac disorders) | 0 (0) | 1 (1)
kidney surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
knee replacement surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
total hip replacement surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
wrist injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
hand and rib injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
torn cartilage in knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Automated Exercise Group (N=52) | Attention Control Group (N=51)
Inury/discomfort (Musculoskeletal and connective tissue disorders) | 8 (8) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes